CLINICAL TRIAL: NCT03836261
Title: A Randomized, Multicenter, Open-Label, Phase 3 Study to Compare the Efficacy and Safety of Acalabrutinib (ACP-196) in Combination With Venetoclax With and Without Obinutuzumab Compared to Investigator's Choice of Chemoimmunotherapy in Subjects With Previously Untreated Chronic Lymphocytic Leukemia Without Del(17p) or TP53 Mutation (AMPLIFY)
Brief Title: Study of Acalabrutinib (ACP-196) in Combination With Venetoclax (ABT-199), With and Without Obinutuzumab (GA101) Versus Chemoimmunotherapy for Previously Untreated CLL
Acronym: AMPLIFY
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Acerta Pharma BV (Industry)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACE-CL-311; D8221C00001 (Other: AstraZeneca); 2023-509349-11-00 (Registry Identifier: CTIS (EU)); 2018-002443-28 (EudraCT Number); NCT05211856 (obsolete NCT alias)
Record Dates: First submitted 2019-02-06; First posted 2019-02-11 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: CLL; Chronic Leukemia Lymphocytic; Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, B-Cell; Leukemia | interventions — acalabrutinib; venetoclax; obinutuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Acalabrutinib, Venetoclax (Experimental): Acalabrutinib in combination with Venetoclax
  Interventions: Drug: Acalabrutinib; Drug: Venetoclax
- Acalabrutinib, Venetoclax, Obinutuzumab (Experimental): Acalabrutinib in combination with Venetoclax with Obinutuzumab
  Interventions: Drug: Acalabrutinib; Drug: Venetoclax; Drug: Obinutuzumab
- Chemoimmunotherapy (Active Comparator): Chemoimmunotherapy
  FCR: Fludarabine, Cyclophosphamide and Rituximab
  BR: Bendamustine and Rituximab
  Interventions: Drug: Chemoimmunotherapy

INTERVENTIONS:
Drug: Acalabrutinib — Acalabrutinib,
  Other Names: Calquence (acalabrutinib)
  Arms: Acalabrutinib, Venetoclax; Acalabrutinib, Venetoclax, Obinutuzumab
Drug: Venetoclax — Venetoclax
  Other Names: Venclyxto, Venclexta
  Arms: Acalabrutinib, Venetoclax; Acalabrutinib, Venetoclax, Obinutuzumab
Drug: Chemoimmunotherapy — fludarabine/cyclophosphamide/rituximab (FCR), bendamustine/rituximab (BR)
  Arms: Chemoimmunotherapy
Drug: Obinutuzumab — Obinutuzumab
  Other Names: Gazyva, Gazyvaro
  Arms: Acalabrutinib, Venetoclax, Obinutuzumab

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of acalabrutinib in combination with venetoclax and acalabrutinib in combination with venetoclax with and without obinutuzumab compared to chemoimmunotherapy in subjects with previously untreated CLL

DETAILED DESCRIPTION:
This randomized, global, multicenter, open-label, Phase 3 study will evaluate the efficacy and safety of AV and AVG versus chemoimmunotherapy (FCR or BR) in subjects with previously untreated CLL without del(17p) or TP53. Subjects will be randomized in a 1:1:1 ratio into 3 arms through a block stratified randomization procedure.

The study includes screening (35 days), treatment (from randomization until study drug discontinuation) and follow-up phase.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ≥18 years of age.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
* Diagnosis of CLL that meets published diagnostic criteria (Hallek et al. 2018)
* Active disease per IWCLL 2018 criteria that requires treatment.
* Participants must use highly effective birth control throughout the study.

Exclusion Criteria:

* Any prior CLL-specific therapies.
* Detected del(17p) or TP53 mutation.
* Transformation of CLL to aggressive non-Hodgkin lymphoma (NHL) (e.g., Richter's transformation, prolymphocytic leukemia [PLL], or diffuse large B cell lymphoma [DLBCL]), or central nervous system (CNS) involvement by leukemia.
* History of confirmed progressive multifocal leukoencephalopathy (PML).
* Received any investigational drug within 30 days before first dose of study drug.
* Major surgical procedure within 30 days before the first dose of study drug.
* Significant cardiovascular disease such as symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of Screening, or any Class 3 or 4 cardiac disease. Note: Subjects with controlled, asymptomatic atrial fibrillation are allowed to enroll on study.
* Malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach, or extensive small bowel resection that is likely to affect absorption, symptomatic inflammatory bowel disease, or partial or complete bowel obstruction, or gastric restrictions and bariatric surgery, such as gastric bypass.
* Received a live virus vaccination within 28 days of first dose of study drug.
* Known history of infection with human immunodeficiency virus (HIV).
* Serologic status reflecting active hepatitis B or C infection.
* History of known hypersensitivity or anaphylactic reactions to study drugs or excipients.
* History of stroke or intracranial hemorrhage within 6 months before first dose of study drug.
* Known bleeding disorders.
* Requires or receiving anticoagulation with warfarin or equivalent vitamin K antagonists.
* Female participants must not be breastfeeding or pregnant.
* Concurrent participation in another therapeutic clinical trial.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 984 (Actual)
Dates: Start 2019-02-25 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate the efficacy of acalabrutinib with venetoclax (Arm A) compared to chemoimmunotherapy fludarabine/cyclophosphamide/rituximab [FCR] or bendamustine/rituximab [BR] (Arm C): PFS | 6 years
  Progression-free survival (PFS) after randomization, defined as the time from randomization to the first occurrence of disease progression or death from any cause (whichever occurs first), as determined by the Independent Review Committee (IRC) according to the International Workshop on Chronic Lymphocytic Leukemia (IWCLL) 2018 criteria

SECONDARY OUTCOMES:
To evaluate the efficacy of acalabrutinib with venetoclax in combination with obinutuzumab (Arm B) compared with FCR or BR (Arm C): PFS | 6 years
  PFS after randomization, defined as the time from randomization to the first occurrence of disease progression or death from any cause (whichever occurs first), as determined by the IRC assessment and investigator assessment
To evaluate the efficacy of acalabrutinib with venetoclax (Arm A) compared with FCR or BR (Arm C): PFS defined the same as above per investigator assessment. | 6 years
  PFS after randomization, defined as the time from randomization to the first occurrence of disease progression or death from any cause (whichever occurs first), as determined by the IRC assessment and investigator assessment

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Brown, Principal Investigator — Dana Farber Mass General Brigham Cancer Care Inc; Barbara Eichhorst, Principal Investigator — Universitätsklinikum Köln; Arnon Kater, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA); Paolo Ghia, Principal Investigator — OSPEDALE S. RAFFAELE - MILANO; John Seymour, Principal Investigator — Peter MacCallum Cancer Ctr
Locations (140):
- United States (15):
  - Research Site, Los Angeles, California
  - Research Site, Redondo Beach, California
  - Research Site, Fort Wayne, Indiana
  - Research Site, Wichita, Kansas
  - Research Site, Louisville, Kentucky
  - Research Site, New Orleans, Louisiana
  - Research Site, Baltimore, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, New York, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Canton, Ohio
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Fort Sam Houston, Texas
  - Research Site, Spokane, Washington
  - Research Site, Tacoma, Washington
- Argentina (3):
  - Research Site, Buenos Aires
  - Research Site, Capital Federal
  - Research Site, Córdoba
- Australia (8):
  - Research Site, Adelaide
  - Research Site, Darlinghurst
  - Research Site, Heidelberg
  - Research Site, Kogarah
  - Research Site, Melbourne
  - Research Site, Nedlands
  - Research Site, Waratah
  - Research Site, Woolloongabba
- Austria (3):
  - Research Site, Krems
  - Research Site, Salzburg
  - Research Site, Vienna
- Brazil (4):
  - Research Site, Goiânia
  - Research Site, Porto Alegre
  - Research Site, Rio de Janeiro
  - Research Site, São Paulo
- Bulgaria (3):
  - Research Site, Plovdiv
  - Research Site, Sofia
  - Research Site, Vratsa
- Canada (7):
  - Research Site, Calgary, Alberta
  - Research Site, Edmonton, Alberta
  - Research Site, Vancouver, British Columbia
  - Research Site, Ottawa, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
- China (16):
  - Research Site, Beijing
  - Research Site, Changchun
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Chongqing
  - Research Site, Guangzhou
  - Research Site, Hangzhou
  - Research Site, Nanchang
  - Research Site, Nanjing
  - Research Site, Shenyang
  - Research Site, Tianjin
  - Research Site, Ürümqi
  - Research Site, Wenzhou
  - Research Site, Wuhan
  - Research Site, Xi'an
  - Research Site, Zhengzhou
- Czechia (6):
  - Research Site, Brno
  - Research Site, Hradec Králové
  - Research Site, Olomouc
  - Research Site, Ostrava - Poruba
  - Research Site, Plzen - Lochotin
  - Research Site, Prague
- Denmark (3):
  - Research Site, Aarhus
  - Research Site, Copenhagen
  - Research Site, Roskilde
- France (6):
  - Research Site, Montpellier
  - Research Site, Paris
  - Research Site, Rennes
  - Research Site, Rouen
  - Research Site, Toulouse
  - Research Site, Villejuif
- Germany (2):
  - Research Site, Paderborn
  - Research Site, Würzburg
- Hungary (3):
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Kaposvár
- Israel (5):
  - Research Site, Haifa
  - Research Site, Jerusalem
  - Research Site, Petah Tikva
  - Research Site, Tel Aviv
  - Research Site, Tel Litwinsky
- Italy (5):
  - Research Site, Meldola
  - Research Site, Milan
  - Research Site, Novara
  - Research Site, Ravenna
  - Research Site, Torino
- Netherlands (5):
  - Research Site, 's-Hertogenbosch
  - Research Site, Almere Stad
  - Research Site, Amsterdam
  - Research Site, Arnhem
  - Research Site, Breda
- Poland (7):
  - Research Site, Brzozów
  - Research Site, Bydgoszcz
  - Research Site, Gdynia
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Lublin
  - Research Site, Wroclaw
- Russia (6):
  - Research Site, Moscow
  - Research Site, Saint Petersburg
  - Research Site, Samara
  - Research Site, Sochi
  - Research Site, Tula
  - Research Site, Volgograd
- Saudi Arabia (3):
  - Research Site, Dammam
  - Research Site, Jeddah
  - Research Site, Riyadh
- Research Site, Bratislava, Slovakia
- South Africa (5):
  - Research Site, Bloemfontein
  - Research Site, Cape Town
  - Research Site, Pretoria
  - Research Site, Randburg
  - Research Site, Soweto
- South Korea (2):
  - Research Site, Incheon
  - Research Site, Seoul
- Spain (7):
  - Research Site, Badalona
  - Research Site, Barcelona
  - Research Site, Madrid
  - Research Site, Majadahonda
  - Research Site, Salamanca
  - Research Site, Santander
  - Research Site, Valencia
- Sweden (3):
  - Research Site, Gothenburg
  - Research Site, Örebro
  - Research Site, Uppsala
- Taiwan (5):
  - Research Site, Kaohsiung City
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
  - Research Site, Taoyuan
- Turkey (Türkiye) (4):
  - Research Site, Ankara
  - Research Site, Izmir
  - Research Site, Kurupelit
  - Research Site, Talas
- United Kingdom (3):
  - Research Site, Cambridge
  - Research Site, Canterbury
  - Research Site, Wolverhampton

REFERENCES:
- [Derived] Brown JR, Seymour JF, Jurczak W, Aw A, Wach M, Illes A, Tedeschi A, Owen C, Skarbnik A, Lysak D, Eom KS, Simkovic M, Pavlovsky MA, Kater AP, Eichhorst B, Miller K, Munugalavadla V, Yu T, de Borja M, Ghia P; AMPLIFY investigators; AMPLIFY Investigators. Fixed-Duration Acalabrutinib Combinations in Untreated Chronic Lymphocytic Leukemia. N Engl J Med. 2025 Feb 20;392(8):748-762. doi: 10.1056/NEJMoa2409804. Epub 2025 Feb 5. PMID 39976417
- [Derived] Alfaifi A, Bahashwan S, Alsaadi M, Ageel AH, Ahmed HH, Fatima K, Malhan H, Qadri I, Almehdar H. Advancements in B-Cell Non-Hodgkin's Lymphoma: From Signaling Pathways to Targeted Therapies. Adv Hematol. 2024 Nov 12;2024:5948170. doi: 10.1155/2024/5948170. eCollection 2024. PMID 39563886
- [Derived] Davids MS, Lampson BL, Tyekucheva S, Wang Z, Lowney JC, Pazienza S, Montegaard J, Patterson V, Weinstock M, Crombie JL, Ng SY, Kim AI, Jacobson CA, LaCasce AS, Armand P, Arnason JE, Fisher DC, Brown JR. Acalabrutinib, venetoclax, and obinutuzumab as frontline treatment for chronic lymphocytic leukaemia: a single-arm, open-label, phase 2 study. Lancet Oncol. 2021 Oct;22(10):1391-1402. doi: 10.1016/S1470-2045(21)00455-1. Epub 2021 Sep 14. PMID 34534514
- [Derived] Gordon MJ, Danilov AV. The evolving role of Bruton's tyrosine kinase inhibitors in chronic lymphocytic leukemia. Ther Adv Hematol. 2021 Jan 30;12:2040620721989588. doi: 10.1177/2040620721989588. eCollection 2021. PMID 33796237